CLINICAL TRIAL: NCT03575754
Title: A Single-center, Feasibility Study to Evaluate the Use and Safety of the Percutaneous Ultrasound Gastrostomy Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CoapTech (Industry)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1801001
Record Dates: First submitted 2018-06-18; First posted 2018-07-03 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Gastrostomy
MeSH Terms: interventions — Gastrostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional (Experimental): This arm utilizes the investigational device, as specified in protocol.
  Interventions: Device: Percutaneous Ultrasound Gastrostomy

INTERVENTIONS:
Device: Percutaneous Ultrasound Gastrostomy — A balloon catheter is inserted into the stomach and used to appose tissue between anterior stomach and skin. Fluid fills the balloon, enabling ultrasound visualization. Then a guidewire is inserted, and pulled out through the mouth to create wire-to-wire (through and through) access. At that point, a gastrostomy tube is placed over it using over-the-wire (push) technique.
  Other Names: Gastrostomy

SUMMARY:
This is a single-center, non-randomized, non-blinded feasibility study to evaluate the performance, safety and tolerability of the Percutaneous Ultrasound Gastrostomy (PUG) procedure that utilizes a novel device in conjunction with widely available ultrasound technology. The procedure will be performed in up to 25 eligible subjects. Patients will be followed for 2 days following performance of PUG to assess for potential complications. If the patient remains hospitalized they will be assessed at date of discharge or Day 30 (whichever is earlier) for potential complications.

DETAILED DESCRIPTION:
Gastrostomy feeding is an established means of delivering adequate nutrition to patients with an inability to meet their metabolic requirements due to inadequate oral intake. Additionally, the gastrostomy tube can be utilized for medication administration in patients unable to otherwise tolerate oral intake. Traditionally, placement of gastrostomy tubes has been performed endoscopically, radiologically or by either laparoscopic or open surgical techniques. More than 200,000 gastrostomy tubes are placed each year in the United States, and that number is expected to increase as the proportion of the population that is elderly grows (Roche et al 2003, Goldberg et al 2005, Lynch et al 2004).

Previous studies have failed to identify a clearly superior technique for placement of feeding tubes (Bravo 2016, Yuan 2016). Percutaneous endoscopic gastrostomy (PEG) was first described by Gauderer et al. in 1980 in a case series of 12 children as an alternative to laparotomy in high-risk patients (Gauderer 1980). There is a high overall success rate of PEG placement at 95-100% (Itkin 2011). Percutaneous endoscopic gastrostomy (PEG) has become the most common method for placement of a gastrostomy tube. This requires the use of specialized equipment and the availability of physicians specifically trained in this procedure. The number of procedures performed yearly to place feeding tubes is expected to rise as the population ages and as some treatments have resulted in some diseases become chronic states rather than invariably fatal conditions.

Challenges to performance of gastrostomy tube placement include the requirement for specialized equipment, specialized areas designated to have this procedure performed as well as the need for proceduralists who are specifically trained in this technique.

The CoapTech device was developed in an effort to reduce the complicated requirements associated with other techniques of gastrostomy placement so that when clinically indicated the procedure can be performed in a safe and timely manner by a wide range of clinicians with various training backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any study-specific assessment is performed
* Male or female ≥18 years of age
* 20≤ BMI ≤30
* Indication for gastrostomy tube placement determined to be present by the primary clinical care team
* Patient determined to be an appropriate candidate for gastrostomy by the study team
* Women of childbearing potential must have negative serum or urine pregnancy test during the current hospitalization

Exclusion Criteria:

* BMI > 30, or BMI < 20
* Temperature ≥ 38 C
* Systolic BP < 100 or > 180 mmHg
* Heart Rate < 50 or > 110
* Presence of a contraindication to being in proximity to a magnet (e.g. pacemaker).
* History of prior gastrostomy, gastrectomy (partial or complete), or abdominal trauma or upper-abdominal surgery.
* Patients with hematocrit <25%, or a history of blood transfusion within the 14 days prior to screening, or active life-threatening GI bleeding.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Involvement in other investigational trials within 30 days prior to screening.
* Any other medical condition(s) that may put the patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study. For example, large or collapsed transverse colon overlapping anterior stomach on pre-existing radiographic scan.
* Anticipated discharge < 36 hours from gastrostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Derived] Accorsi F, Chung J, Mujoomdar A, Wiseman D, Kribs S, Cool DW. Percutaneous ultrasound gastrostomy (PUG): first prospective clinical trial. Abdom Radiol (NY). 2021 Nov;46(11):5377-5385. doi: 10.1007/s00261-021-03200-x. Epub 2021 Jul 9. PMID 34240242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began Oct 2018 and concluded Apr 2020. Patients referred to Interventional Radiology for gastrostomy tube placement were approached for consent at least 24hrs pre-procedure in clinic or in hospital. When patients lacked capacity to consent, a surrogate decision maker was approached or reached remotely for telephone consent.
Pre-assignment Details: No pre-assignment methods were employed in this protocol
Groups:
- Prospective PUG Cohort: Patients meeting all the inclusion criteria and none of the exclusion criteria and provided study consent who received the Percutaneous Ultrasound Gastrostomy (PUG) procedure
- Matched Retrospective RIG Cohort: Patients who previously received the standard of care Radiologic Inserted Gastrostomy (RIG) procedure. A waiver of consent was provided by the Research Ethics Board for this study arm.
Period: Overall Study
Arm/Group | Prospective PUG Cohort | Matched Retrospective RIG Cohort
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional | Matched Retrospective RIG Cohort | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (15) | 66 (14) | 65 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 23 | 23 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 21 | 0 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 25 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Device Related Adverse Events
Description: the number of enrolled subjects who have a serious, adverse event during placement of a gastrostomy tube using the PUG procedure. Adverse events were defined by the Clavien-Dindo classification system of surgical complications. For the purpose of this study, minor adverse events are defined as Grade I-II and serious adverse events as Grade III-V. See references for relevant citation.
Time Frame: Discharge or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective PUG Cohort | Matched Retrospective RIG Cohort
Number analyzed (Participants) | 25 | 25
Participants | 1 | 5

2. Secondary Outcome: Severity of Serious Device Related Adverse Events
Description: the severity of any serious, device-related adverse event during placement of a gastrostomy tube using the PUG procedure (if applicable). Adverse events were defined by the Clavien-Dindo classification system of surgical complications. For the purpose of this study, minor adverse events are defined as Grade I-II and serious adverse events as Grade III-V. See references for relevant citation.
Time Frame: Discharge or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective PUG Cohort | Matched Retrospective RIG Cohort
Number analyzed (Participants) | 25 | 25
Participants
  Grade IIIA: Complications requiring surgical, endoscopic or radiological intervention w/o anesthesia | 1 | 5
  Grade IIIB: Complications requiring surgical, endoscopic or radiological intervention w anesthesia | 0 | 0
  Grade IV: Life-threatening complications | 0 | 0
  Grade V: Death of patient | 0 | 0

3. Secondary Outcome: Number of Participants With Technically Successful Gastrostomy Tube Placement
Description: the number of enrolled subjects who have successful placement of a gastrostomy tube
Time Frame: Discharge or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective PUG Cohort | Matched Retrospective RIG Cohort
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

4. Secondary Outcome: Length of Angiographic Suite Usage
Description: Length of angiographic suite usage in minutes
Time Frame: Discharge or 30 days
Population: 22 of the participants in the Prospective PUG Cohort and 25 participants in the Matched Retrospective RIG Cohort were analyzed in this group as each received gastrostomy procedure within the Angiosuite. 3 participants in the Prospective PUG Cohort were excluded in this analysis as procedures were performed at the bedside on the Intensive Care Unit (ICU).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Prospective PUG Cohort | Matched Retrospective RIG Cohort
Number analyzed (Participants) | 22 | 25
minutes | 68 (24.5) | 39.3 (15)

ADVERSE EVENTS:
Time Frame: At least 48hrs post-procedure until discharge from hospital or 30 days post-procedure (whichever came sooner)
Description: All cause adverse events observed in study participants were defined by the Clavien-Dindo classification system of surgical complications. For the purpose of this study, minor adverse events are defined as Grade I-II and major adverse events as Grade III-V.
Arm/Group | Prospective PUG Cohort | Matched Retrospective RIG Cohort
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 5/25
Other Adverse Events (participants affected / at risk) | 3/25 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective PUG Cohort (N=25) | Matched Retrospective RIG Cohort (N=25)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrostomy Tube Failure (Gastrointestinal disorders) | 0 (0) | 5 (5) — Gastrostomy tube failure requiring non-invasive or surgical intervention to replace
Abdominal Wall Abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective PUG Cohort (N=25) | Matched Retrospective RIG Cohort (N=25)
Mild Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Local Stomal Site Infection (Infections and infestations) | 2 (2) | 0 (0) — Infection seeded at the site of the gastrostomy tube tract

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03575754/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03575754/SAP_001.pdf